CLINICAL TRIAL: NCT06908668
Title: A Prospective, Multicenter, Randomized Controlled Phase II Study to Evaluate the Efficacy and Safety of Adebrelimab Combined With Chemotherapy With or Without Radiotherapy as Neoadjuvant Treatment for HER2-Negative Locally Advanced Breast Cancer
Brief Title: Evaluate the Efficacy and Safety of Adebrelimab Combined With Chemotherapy With or Without Radiotherapy as Neoadjuvant Treatment for HER2-Negative Locally Advanced Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Deputy Director, Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC5177
Record Dates: First submitted 2025-03-18; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: HER2-Negative Locally Advanced Breast Cancer
MeSH Terms: interventions — Immunotherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant Chemotherapy Combined with Immunotherapy and Radiotherapy (Experimental): 1. Recommended Chemotherapy Regimen and Doses:
     Albumin-bound Paclitaxel 260 mg/m² on Day 1, every 3 weeks (Q3W) × 4 cycles, followed by Epirubicin 90 mg/m² on Day 1 + Cyclophosphamide 600 mg/m² on Day 1, every 3 weeks (Q3W) × 4 cycles.
  2. Recommended Immunotherapy Dose:
     Adebrelimab 1200 mg, repeated every 3 weeks, starting simultaneously with neoadjuvant chemotherapy and continuing for 1 year (including postoperative administration).
  3. Radiotherapy:
  Preoperative Radiotherapy:
  Positioning: Immobilization with a neck-chest integrated frame, combined CT and MRI positioning with image fusion. Diagnostic MRI images can also be fused simultaneously. CT positioning should be performed with a plain scan, with a slice thickness of 3 mm. MRI positioning should include at least three sequences: T1-enhanced, T2 fat-suppressed, and DWI.
  Target and Normal Organ Contouring:
  GTVp (Gross Tumor Volume - Primary): Define the breast tumor target area based on MRI, CT, physical examination, and ultrasoun
  Interventions: Drug: Neoadjuvant Chemotherapy Combined with Immunotherapy and Radiotherapy
- Neoadjuvant Chemotherapy Combined with Immunotherapy (Active Comparator): 1. Recommended Chemotherapy Regimen and Doses:
     Albumin-bound Paclitaxel 260 mg/m² on Day 1, every 3 weeks (Q3W) × 4 cycles, followed by Epirubicin 90 mg/m² on Day 1 + Cyclophosphamide 600 mg/m² on Day 1, every 3 weeks (Q3W) × 4 cycles.
  2. Recommended Immunotherapy Dose:
  Adebrelimab 1200 mg, repeated every 3 weeks, starting simultaneously with neoadjuvant chemotherapy and continuing for 1 year (including postoperative administration).
  Interventions: Drug: Neoadjuvant Chemotherapy Combined with Immunotherapy

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy Combined with Immunotherapy and Radiotherapy — 1. Recommended Chemotherapy Regimen and Doses:
     Albumin-bound Paclitaxel 260 mg/m² on Day 1, every 3 weeks (Q3W) × 4 cycles, followed by Epirubicin 90 mg/m² on Day 1 + Cyclophosphamide 600 mg/m² on Day 1, every 3 weeks (Q3W) × 4 cycles.
  2. Recommended Immunotherapy Dose:
     Adebrelimab 1200 mg, repeated every 3 weeks, starting simultaneously with neoadjuvant chemotherapy and continuing for 1 year (including postoperative administration).
  3. Radiotherapy:
  Preoperative Radiotherapy:
  Positioning: Immobilization with a neck-chest integrated frame, combined CT and MRI positioning with image fusion. Diagnostic MRI images can also be fused simultaneously. CT positioning should be performed with a plain scan, with a slice thickness of 3 mm. MRI positioning should include at least three sequences: T1-enhanced, T2 fat-suppressed, and DWI.
  Target and Normal Organ Contouring:
  GTVp (Gross Tumor Volume - Primary): Define the breast tumor target area based on MRI, CT, physical examination, and ultrasound
  Arms: Neoadjuvant Chemotherapy Combined with Immunotherapy and Radiotherapy
Drug: Neoadjuvant Chemotherapy Combined with Immunotherapy — 1. Recommended Chemotherapy Regimen and Doses:
     Albumin-bound Paclitaxel 260 mg/m² on Day 1, every 3 weeks (Q3W) × 4 cycles, followed by Epirubicin 90 mg/m² on Day 1 + Cyclophosphamide 600 mg/m² on Day 1, every 3 weeks (Q3W) × 4 cycles.
  2. Recommended Immunotherapy Dose:
  Adebrelimab 1200 mg, repeated every 3 weeks, starting simultaneously with neoadjuvant chemotherapy and continuing for 1 year (including postoperative administration).
  Arms: Neoadjuvant Chemotherapy Combined with Immunotherapy

SUMMARY:
A Prospective, Multicenter, Randomized Controlled Phase II Study to Evaluate the Efficacy and Safety of Adebrelimab Combined with Chemotherapy with or without Radiotherapy as Neoadjuvant Treatment for HER2-Negative Locally Advanced Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged between 18 and 70 years old.
2. Pathologically confirmed as invasive breast cancer, with immunohistochemical staining indicating HER2 negativity, as specifically referenced in the guidelines of the American Society of Clinical
3. Oncology/College of American Pathologists (ASCO/CAP).
4. Clinical stage II-III, patients who are planned to undergo neoadjuvant treatment to downstage for surgery or who wish to have breast-conserving surgery after neoadjuvant treatment.
5. The breast tumor is suitable for SBRT (stereotactic body radiotherapy) (tumor distance from the skin > 5 mm, without invasion of the ribs or intercostal muscles).
6. No distant metastasis detected by clinical examination combined with imaging studies (including but not limited to liver ultrasound, chest CT, bone scan, PET-CT).
7. Adequate organ function (hemoglobin ≥ 100 g/L, white blood cells ≥ 3×10⁹/L, neutrophils ≥ 1.5×10⁹/L, platelets ≥ 80×10⁹/L; creatinine ≤ 132 μmol/L; alanine aminotransferase/aspartate aminotransferase ≤ 2.5×upper normal limit [UNL]).
8. Capable of undergoing breast magnetic resonance imaging (MRI) scans. Eligible for follow-up conditions.
9. The subject is able to sign the informed consent form to participate in the study.
10. Women of childbearing age are not pregnant, not breastfeeding, and are using effective contraception.

Exclusion Criteria:

1. Prior receipt of chest radiotherapy, chemotherapy, or immunotherapy.
2. History of other malignancies, with the exception of adequately treated basal cell carcinoma of the skin, carcinoma in situ of the cervix, or papillary thyroid cancer.
3. Patients with active fibroconnective tissue diseases, risk of active autoimmune diseases, or a history of autoimmune diseases that may involve the central nervous system, including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener's syndrome, granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, autoimmune hepatitis, systemic sclerosis, Hashimoto's thyroiditis, autoimmune vasculitis, and autoimmune neuropathies (e.g., Guillain-Barré syndrome). The following exceptions apply: Type I diabetes mellitus, stable hypothyroidism on hormone replacement therapy (including hypothyroidism due to autoimmune thyroid disease), psoriasis or vitiligo not requiring systemic therapy, and autoimmune diseases caused by B cells or anti-self-antigen antibodies.
4. Pulmonary disease defined as ≥ Grade 3 according to the NCI-CTCAE v5.0; history of interstitial lung disease (ILD) requiring corticosteroid treatment (including pulmonary fibrosis or radiation pneumonitis), or current ILD or ≥ Grade 2 radiation pneumonitis.
5. Severe comorbidities or active diseases:

   a) History of severe cardiovascular and cerebrovascular diseases, including but not limited to: i. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, or third-degree atrioventricular block; ii. QT interval prolongation at rest (QTc > 450 msec in males or > 470 msec in females); iii. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other Grade 3 or higher cardiovascular and cerebrovascular events within 6 months prior to the first dose; iv. Presence of heart failure with New York Heart Association (NYHA) functional class ≥ II.

   b) Poorly controlled diabetes for > 1 month: fasting blood glucose > 10 mmol/L, or postprandial 2-hour blood glucose > 13 mmol/L.

   c) Poorly controlled psychiatric disorders with an episode or exacerbation within the past 6 months.

   d) Active infection. e) Positive for human immunodeficiency virus (HIV) antibodies. Other diseases that are not suitable for immunotherapy, or a history of other malignancies.
6. Presence of severe internal medical conditions that may affect radiotherapy or immunotherapy.
7. Pregnant or breastfeeding women.
8. History of allergy to components of radiotherapy or immunotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2028-09-10 (Estimated); Study Completion 2028-09-10 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | 24 months
  For binary efficacy endpoints (including pCR, ORR, etc.), the number of subjects and percentage in each category will be summarized, and the 95% confidence interval for the rate will be calculated using the Clopper-Pearson method.